CLINICAL TRIAL: NCT07012525
Title: Clinical Evaluation of Photobiomodulated Hyaluronic Acid Therapy for Interdental Papillary Loss: Minimal Invasive Blind Split Mouth Technique
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dar Al Uloom University (Other)
Responsible Party: Principal Investigator, Sally Abd-ElMeniem ElHaddad, Assist. Prof. Periodontology and Oral Medicine, Dar Al Uloom University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31-05-2024
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Interdental Papillae Reconstruction
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Study Type: Interventional (Clinical Trial) Model: Split-Mouth, Parallel Assignment Masking: Single-Blind (Outcomes Assessor) Primary Purpose: Treatment This study follows a split-mouth randomized controlled design, where each participant serves as their own control. The oral cavity is divided into right and left maxillary quadrants. One quadrant (control group) will receive hyaluronic acid (HA) filler only, while the other quadrant (experimental group) will receive HA filler combined with photobiomodulation therapy (PBMT).
  This within-subject model minimizes inter-individual variability and allows for more accurate comparison of treatment efficacy between the two modalities. Randomization determines which side receives the PBMT-enhanced therapy. Outcome assessors are blinded to group allocation to reduce bias during follow-up measurements.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photobiomodulation + Hyaluronic Acid (Experimental): This arm includes the test sites (e.g., left maxillary quadrant) in each participant. The same dose of hyaluronic acid (0.2 mL of 0.8% gel) will be injected in the same manner as in the control group. However, photobiomodulation therapy (PBMT) using a diode laser (wavelength 630-670 nm, 25 mW, 1.875 J/cm² for 20 seconds) will be applied before and after the injection. Laser application will be repeated at every follow-up appointment to promote tissue healing, angiogenesis, and papillary regeneration.
  Interventions: Procedure: Photobiomodulation Therapy + Hyaluronic Acid Gel Injection
- Hyaluronic Acid Gel Injection only (Active Comparator): This arm includes the control sites (e.g., right maxillary quadrant) in each participant. The interdental papilla with Class I deficiency will be treated using 0.2 mL of 0.8% commercial hyaluronic acid gel, injected 2-3 mm apical to the papilla tip. This is a commonly used non-surgical soft tissue filler in periodontal and esthetic procedures. No photobiomodulation therapy will be applied in this arm.
  Interventions: Drug: Hyaluronic Acid Gel Injection

INTERVENTIONS:
Procedure: Photobiomodulation Therapy + Hyaluronic Acid Gel Injection — This arm includes the test sites (e.g., left maxillary quadrant) in each participant. The same dose of hyaluronic acid (0.2 mL of 0.8% gel) will be injected in the same manner as in the control group. However, photobiomodulation therapy (PBMT) using a diode laser (wavelength 630-670 nm, 25 mW, 1.875 J/cm² for 20 seconds) will be applied before and after the injection. Laser application will be repeated at every follow-up appointment to promote tissue healing, angiogenesis, and papillary regeneration.
  Arms: Photobiomodulation + Hyaluronic Acid
Drug: Hyaluronic Acid Gel Injection — This arm includes the control sites (e.g., right maxillary quadrant) in each participant. The interdental papilla with Class I deficiency will be treated using 0.2 mL of 0.8% commercial hyaluronic acid gel, injected 2-3 mm apical to the papilla tip. This is a commonly used non-surgical soft tissue filler in periodontal and esthetic procedures. No photobiomodulation therapy will be applied in this arm.
  Arms: Hyaluronic Acid Gel Injection only

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a minimally invasive therapy combining photobiomodulation (PBMT) with injectable dermal filler (hyaluronic acid) in adult patients (ages 20-40) with interdental papillary loss (Norland & Tarnow Class I) in the maxillary anterior region.

The main questions it aims to answer are:

Does PBMT enhance the regenerative effect of hyaluronic acid filler in restoring the interdental papilla? Is the combined therapy superior to dermal filler alone in achieving long-term aesthetic and clinical stability?

Researchers will compare:

Group I (control) - hyaluronic acid filler alone vs. Group II (experimental) - PBMT applied before and after hyaluronic acid filler to see if PBMT contributes to better papilla height, width, and volume restoration over 12 months.

Participants will:

Undergo standard periodontal cleaning and education 4 weeks before treatment Receive local anesthesia and dermal filler injections in both quadrants (split-mouth design)

Have PBMT applied in one quadrant only (Group II) Be followed up at regular intervals (1 week to 12 months) for clinical measurements and digital image analysis of papilla dimensions This study introduces a non-surgical, patient-friendly technique that may enhance soft tissue regeneration in esthetic areas, offering a potential breakthrough in managing interdental papillary loss.

DETAILED DESCRIPTION:
This study explores a novel, minimally invasive therapeutic approach to treating interdental papillary loss (IDP)-a condition with both functional and esthetic consequences, particularly in the maxillary anterior region. While surgical techniques for papilla regeneration have been investigated for decades, success has been limited due to anatomical challenges such as restricted blood supply and the small volume of tissue involved. Additionally, many of these procedures are invasive, complex, and do not guarantee long-term stability.

The proposed study evaluates the synergistic effect of photobiomodulation therapy (PBMT), formerly known as low-level laser therapy (LLLT), when combined with injectable hyaluronic acid (HA) dermal filler. PBMT is known to enhance microcirculation, stimulate fibroblast activity, and promote angiogenesis, all of which may contribute to improved tissue regeneration. HA, on the other hand, supports extracellular matrix remodeling, tissue hydration, and wound healing. While HA has shown some promise when used alone for papilla reconstruction, recurrence of papillary loss has been reported within 6-12 months post-treatment.

This clinical trial employs a split-mouth, randomized controlled design to compare two interventions within the same patient-HA filler alone versus HA combined with PBMT. By minimizing inter-patient variability, this design enhances internal validity and provides a more reliable comparison of treatment efficacy.

Throughout a 12-month follow-up period, the study will assess changes in papillary height, width, and overall tissue volume using standardized clinical measurements and digital imaging analysis. Additionally, the PBMT group will receive laser therapy at each follow-up session to evaluate its ongoing regenerative contribution.

This study aims to introduce a patient-friendly, conservative alternative to surgical procedures, with the potential to become a predictable and reproducible technique in the esthetic zone. If successful, it may offer a paradigm shift in managing one of the most challenging soft tissue defects in periodontal and esthetic dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 40 years
* Presence of at least two non-adjacent interdental papilla defects (Class I, Norland & Tarnow classification) in the maxillary anterior region
* Healthy periodontal status, with:
* Probing depth ≤ 3 mm
* No gingival recession
* No tooth mobility (Score 0)
* No interdental bone loss on radiographs
* Non-smokers
* No previous orthodontic treatment
* Free from gingival or dental surface alterations (e.g., abfraction, irregularities, or overcontouring)
* Systemically healthy (no systemic diseases or conditions affecting healing or immune function)
* Willing and able to comply with study procedures and follow-up visits
* Provided written informed consent after explanation of study procedures

Exclusion Criteria:

* Candidates will be excluded if they meet any of the following:
* Systemic diseases or medications known to affect soft tissue healing (e.g., diabetes, immunosuppressants)
* Pregnancy or lactation
* History of periodontal surgery in the study area
* Known allergy or hypersensitivity to hyaluronic acid or local anesthetics
* Current use of anti-inflammatory drugs, anticoagulants, or antibiotics that could affect healing
* Poor oral hygiene or non-compliance during pre-treatment phase
* Participation in another clinical trial within the last 3 months

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Papillary Deficient Area | Baseline, 1 month, 3 months, 6 months, and 12 months
  This outcome measures the change in the total area of interdental papillary deficiency (in mm²), calculated using standardized measurements of papillary height and width. The area is estimated using the formula:
  Area = ½ × Papillary Width × Papillary Deficient Height.
  Method of Assessment:
  Clinical measurements with a UNC-15 probe and digital photographic analysis.

SECONDARY OUTCOMES:
Change in Papillary Width | Baseline and follow-up at 1, 3, 6, and 12 months
  Measures the horizontal base width of the interdental papilla at the crestal level between adjacent teeth.
  Assessment Tool:
  Clinical probing and digital image analysis.
Change in Papillary Deficient Height | Baseline and follow-up at 1, 3, 6, and 12 months
  Vertical distance (in mm) from the tip of the papilla to the contact point between adjacent teeth.
  Assessment Tool:
  Periodontal probe (UNC-15) and digital images.
Digital Image Analysis Score | Baseline and follow-up at 1, 3, 6, and 12 months
  Quantitative assessment of papillary volume and soft tissue contour using standardized intraoral photographs and imaging software.
Patient Satisfaction and Aesthetic Score | At 3, 6, and 12 months
  Patient-reported outcomes evaluating satisfaction with esthetics and comfort using a visual analog scale (VAS) from 0 to 10.
Incidence of Adverse Effects | throughout the study duration (from initial treatment up to 12 months)
  Monitors for soft tissue reactions, pain, inflammation, or infection at treatment sites.

CONTACTS AND LOCATIONS:
Overall Officials: SREIC College of dentistry, Dar AlUloom University, Study Director — College of Dentistry, Dar AlUloom University, SA
Locations (1):
- College of Dentistry, Dar AlUloom University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Demographic data: age, sex, and quadrant assignment (test vs. control)
  Papillary measurements:
  Papillary width
  Papillary deficient height
  Calculated deficient area (mm²)
  Digital image analysis scores: baseline and all follow-up intervals
  Patient-reported outcomes: aesthetic satisfaction scores (VAS)
  Adverse events: type, frequency, and severity of any reported reactions
  All data will be anonymized to ensure participant confidentiality in accordance with applicable ethical and legal standards.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Start Date:
  Six months after publication of the primary study results in a peer-reviewed journal.
  End Date:
  Five years from the IPD availability start date.